CLINICAL TRIAL: NCT03256097
Title: Voice Guard Processing Evaluation in a Cohort of Subjects Implanted With the Neuro Cochlear Implant System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PIC_12
Record Dates: First submitted 2017-08-14; First posted 2017-08-21 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Cochlear Implantation
Keywords: Sound processing strategy

STUDY DESIGN:
Intervention Model Description: A-B-A vs B-A-B
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XDP - VG - XDP (Experimental): order of testing: XDP - VG - XDP
  Interventions: Device: XDP sound processing strategy - Period 0; Device: XDP sound processing strategy - Period 1; Device: VG sound processing strategy - Period 2; Device: XDP sound processing strategy - Period 3; Device: Voice Track
- VG - XDP - VG (Experimental): order of testing: VG - XDP - VG
  Interventions: Device: XDP sound processing strategy - Period 0; Device: VG sound processing strategy - Period 1; Device: XDP sound processing strategy - Period 2; Device: VG sound processing strategy - Period 3; Device: Voice Track

INTERVENTIONS:
Device: XDP sound processing strategy - Period 0 — XDP is a cochlear implant sound processing strategy that coverts environmental sound into meaningful information that a cochlear implant users' brain can comprehend.
Device: XDP sound processing strategy - Period 1 — XDP is a cochlear implant sound processing strategy that coverts environmental sound into meaningful information that a cochlear implant users' brain can comprehend.
  Arms: XDP - VG - XDP
Device: VG sound processing strategy - Period 1 — Voice Guard is a cochlear implant sound processing strategy that coverts environmental sound into meaningful information that a cochlear implant users' brain can comprehend.
  Arms: VG - XDP - VG
Device: XDP sound processing strategy - Period 2 — XDP is a cochlear implant sound processing strategy that coverts environmental sound into meaningful information that a cochlear implant users' brain can comprehend.
  Arms: VG - XDP - VG
Device: VG sound processing strategy - Period 2 — Voice Guard is a cochlear implant sound processing strategy that coverts environmental sound into meaningful information that a cochlear implant users' brain can comprehend
  Arms: XDP - VG - XDP
Device: XDP sound processing strategy - Period 3 — XDP is a cochlear implant sound processing strategy that coverts environmental sound into meaningful information that a cochlear implant users' brain can comprehend.
  Arms: XDP - VG - XDP
Device: VG sound processing strategy - Period 3 — Voice Guard is a cochlear implant sound processing strategy that coverts environmental sound into meaningful information that a cochlear implant users' brain can comprehend
  Arms: VG - XDP - VG
Device: Voice Track — Voice Track is a cochlear implant noise cancellation system which is designed to reduce the adverse effect of background noise on speech perception through cochlear implants

SUMMARY:
The study aims to compare two different cochlear implant sound processing strategies. All the participants will start off with a sound processing strategy called the XDP (extended performance). At the 3 month stage, half of the participants would randomly be selected and offered a sound processing strategy called the Voice Guard. Following that, the sound processing strategies will be altered and evaluated every 3 months at the 6th, 9th and 12th month of cochlear implant use.

DETAILED DESCRIPTION:
Voice Guard and XDP are two different cochlear implant sound processing strategies. The Voice Guard sound coding strategy is adaptive in nature and can alter the output from the cochlear implant based on the levels of the listening environment. Hence, it can adapt to soft, medium or conversational and loud speech levels.The XDP on the other hand is not adaptive and cannot alter the cochlear implant output according to the levels of the listening environment.

In the study we are hypothesising that the Voice Guard sound processing strategy will perform better than the XDP strategy for soft (40 dB SPL) and loud (85 dB SPL) speech input levels. Speech perception scores will be recorded at 40, 65 and 85 dB SPL and a cross over study design has been adopted.

In addition, the efficacy of a cochlear implant sound reduction technique called Voice Track will also be evaluated. The Voice Track is designed to reduce the adverse effect of background noise on cochlear implant speech perception.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 70 years
* Individuals with post-lingual hearing loss
* Individuals with no language and speech production disorders
* Individuals who are native speakers of English
* Individuals meeting NICE candidacy criteria for CI surgery
* Individuals undergoing primary unilateral cochlear implantation

Exclusion Criteria:

* Medical conditions contraindicating CI surgery
* Individuals with anatomical anomalies of the auditory system
* Individuals with additional mental health issues or and/or cognitive impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Speech perception scores in quite and in noise | 12 months
  Speech perception with each intervention will be measured and a score between 0 to 100% will be obtained

SECONDARY OUTCOMES:
Patient reported outcome measure | 12 months
  Glasgow Hearing aid Benefit profile will be administered to assess patient reported benefit with each intervention

CONTACTS AND LOCATIONS:
Overall Officials: James Tysome, Principal Investigator — Consultant Head and Neck Surgeon, Addenbrookes Hospital
Locations (2):
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge University Hospitals Trust, Cambridge, Cambridgeshire
  - Queen Elizabeth Hospital, University of Birmingham NHS Hospitals Trust, Birmingham, West Midlands